CLINICAL TRIAL: NCT04842734
Title: Comparison of the Effect of Online Physical Exercise and Computerized Cognitive Stimulation in Patients With Alzheimer's Disease During the Covid-19 Pandemic
Brief Title: Comparison of the Effect of Online Physical Exercise and Computerized Cognitive Stimulation in Patients With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Ebru Akbuğa Koç, Lecturer, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25.03.2021/37
Record Dates: First submitted 2021-04-10; First posted 2021-04-13 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease; Telerehabilitation; Online Physical Exercise; Computerized Cognitive Stimulation; Covid-19 Pandemic
Keywords: Alzheimer's disease; Telerehabilitation; Physical exercise; Computerized Cognitive Stimulation; Covid-19 Pandemic; Cognitive Stimulation; Online physical exercise; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease; COVID-19; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: It is planned to include 60 individuals diagnosed with AD according to DSM-IV diagnostic criteria by the neurologist. Individuals will be randomly divided into three groups; as the physical exercise group (n=20), physical exercise and cognitive stimulation (n=20) and the control group (n=20) according to inclusion criteria
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical exercise and computerized cognitive stimulation (Experimental): Supervised Physical Exercise Program (SPEP) sessions will be performed simultaneously online together with the physiotherapist and the patient. Participants will be able to do the exercises together with their caregivers if needed.
  The Computerized Cognitive Stimulation Program (CCSP) (Beynex) will be planned for 12 weeks, 5 days a week, approximately 10 minutes, for a total of 40 sessions.
  Fisrtly, the use of CCSP will be demonstrated to the patients. Then, it will be given as home program. While the patients play the games in CCSP via their smartphones, their caregivers will be informed in detail about accompanying the patients if they need it. The follow-up of cognitive stimulation will be made with the person accompanying the patient over the phone.
  Individuals will be evaluated by a physiotherapist who will perform the assessment at pre-treatment, post-treatment (12th week) and follow-up period (24th week).
  Interventions: Other: Physical exercise and computerized cognitive training
- physical exercise (Experimental): SPEP sessions will be demonstrated to individuals by a 6-year-experienced physiotherapist via videoconference (Zoom Inc.) and the exercises will be performed simultaneously online together with the physiotherapist and the patient. Participants will be able to do the exercises together with their caregivers if needed.
  Individuals will be evaluated by a physiotherapist who will perform the assessment at pre-treatment, post-treatment (12th week) and follow-up period (24th week).
  Interventions: Other: Physical exercise
- control (No Intervention): The individuals included in this group will be informed that they should continue their normal daily life activities.
  Individuals will be evaluated by a physiotherapist who will perform the assessment at pre-treatment, post-treatment (12th week) and follow-up period (24th week).

INTERVENTIONS:
Other: Physical exercise — SPEP are planned for 12 weeks, 2 times a week, once a day, 60 minutes / 1 hour
  Arms: physical exercise
Other: Physical exercise and computerized cognitive training — SPEP are planned for 12 weeks, 2 times a week, once a day, 60 minutes / 1 hour. The CCSP is planned for 12 weeks, minimum 3 to maximum 5 days a week, approximately 10 minutes, for a total of 36-60 sessions
  Arms: Physical exercise and computerized cognitive stimulation

SUMMARY:
Our aim has been determined to investigate the effect of physical exercise alone and in combination with cognitive exercise, on cognitive, physical function and quality of life in individuals with Alzheimer's Disease during the Covid-19 pandemic period.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years and older
* Diagnosed with AD according to DSM-IV diagnostic criteria by a neurologist,
* MOCA ≥ 13
* Clinical Dementia Rating Scale < 2
* Having sufficient wireless support or telephone connection where the person lives
* Who gave consent to participate in the study
* No history of any neurological or orthopedic injury that could prevent participation in the study and affect functional mobility.

Exclusion Criteria:

* Geriatric Depression Scale score > 11
* Various mobility restrictions, musculoskeletal disorders, (wheelchair use, etc.)
* Clinically significant aphasia (must be able to understand the therapist's commands)
* Significant visual or sensory impairment
* MoCA < 13
* Having a severe musculoskeletal disorder
* Having paralysis
* Impaired balance
* The presence of severe lung and heart disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Related Quality of Life Scale | 24 weeks
  This scale evaluates health-related quality of life in individuals with AD. The scale includes 40 questions in total and examines 5 quality of life domains (A-Social Interaction, B-Self Awareness, C-Affect and Mood, D- Enjoying Activities, E-Interaction with the Environment).
Montreal Cognitive Assessment Scale | 24 weeks
  MOCA is a short cognitive assessment method developed to detect particularly mild stages of cognitive impairment.
Berg Balance Scale | 24 weeks
  Berg Balance Scale measures static and dynamic balance in elderly individuals.
Time up and Go Test | 24 weeks
  TUG test evaluates fall risk, mobility and physical performance in the elderly
Sit to Stand Test | 24 weeks
  Sit-to-stand test will be performed on an armless chair with a height of 46 cm to determine the physical fitness level of elderly individuals
Arm Curl Test | 24 weeks
  The Arm Curl test is one of the subtests of the Senior fitness test and it is performed to evaluate upper extremity muscle strength

SECONDARY OUTCOMES:
Katz Activities of Daily Living Scale | 24 weeks
  Katz ADLs consist of six questions that include information about bathing, dressing, toilet, movement, excretion, and feeding activities.
Lawton Instrumental Activities of Daily Living Scale | 24 weeks
  Lawton IADL scale consists of 8 items and a single subscale. In addition, it consists of eight questions about using the phone, preparing meals, shopping, doing daily household chores, washing clothes, getting on the transportation vehicle, taking medicines and money management
Geriatric Depression Scale (Short Form) | 24 weeks
  The GDS Short Form (GDS-15) is a 15-item scale that is used for the diagnosis of depression in elderly individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided